CLINICAL TRIAL: NCT01801319
Title: A Clinical Evaluation of Subcallosal Cingulate Gyrus Deep Brain Stimulation for Treatment-Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-08-07; Health Canada 148956 (Other: Health Canada)
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Treatment Resistant Depression; Depressive Disorder
Keywords: major depressive disorder (MDD); deep brain stimulation (DBS); subcallosal cingulate gyrus; Therapy-Resistant Depression; Electrical Stimulation of the Brain; Brain Stimulation, Deep
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulation (Active Comparator): Libra Deep Brain Stimulation System is implanted and activated post implantation
  Interventions: Device: Libra Deep Brain Stimulation System
- No Stimulation (Sham Comparator): The Libra DBS System is implanted and not activated
  Interventions: Device: Libra Deep Brain Stimulation System

INTERVENTIONS:
Device: Libra Deep Brain Stimulation System

SUMMARY:
This is a randomized, placebo-controlled double-blind cross-over trial evaluating the safety, efficacy, daily functioning, and health-related quality of life of Subcallosal Cingulate Gyrus Deep Brain Stimulation (SCG DBS) for participants with Treatment-Resistant Depression (TRD). A total of 40 eligible participants will be randomized to four treatment sequences (10 participants per sequence). Each participant will be treated over a 6-month period with active or sham stimulation in which both the participants and the attending psychiatrists will be blinded to treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (non-pregnant) ages 21-70 years;
2. Diagnosed with non-psychotic major depressive disorder, single or recurrent episode by DSM-IV-TR criteria;
3. First episode onset before age 45;
4. Current episode > 12 months duration;
5. In the current episode: Documented resistance (i.e. persistence of the major depressive episode) to a minimum of 4 adequate depression treatments from at least 3 different treatment categories (e.g. SSRI's, SNRI's, TCA's, MAO-inhibitors, Mirtazipine, Nefazodone, Trazodone, Bupropion, lithium augmentation, thyroid augmentation, ECT); Adequacy of treatments as defined by a score of at least 3 according to the amended Antidepressant Treatment History Form (ATHF) criteria;
6. Hamilton Depression Rating Scale (HDRS) of > 20 at 3 separate baseline visits, rated by 2 separate psychiatrists, Baseline 2 and Baseline 3 HDRS scores cannot improve ≥ 25%;

Exclusion Criteria:

1. A diagnosis of a bipolar I or bipolar II disorder by DSM-IV-TR criteria;
2. Meets criteria for borderline or antisocial personality disorder in the last 12 months by DSM-IV-TR criteria, derived from the Cluster B Personality.
3. In the current depressive episode, has been diagnosed with General Anxiety Disorder (GAD) - as defined by the DSM-IV-TR, and GAD is the primary diagnosis;
4. Has an intracranial Central Nervous System (CNS) disease that impairs motor, sensory or cognitive function or that requires intermittent or chronic medication (e.g., Parkinson's Disease, migraine, stroke, Huntington's, head trauma, etc.) with exception to non-migraine headaches;
5. Has been diagnosed with fibromyalgia or has a current condition which requires chronic pain narcotic usage (e.g. morphine, methadone);
6. Has been currently diagnosed with chronic fatigue syndrome;
7. Substantial suicidal risk as defined by (1) a current plan and intent, (2) clinician judgment that there is a clear immediate intent for self-harm, (3) more than 3 suicide attempts within the last 12 months;
8. Co-morbid obsessive compulsive disorder, post-traumatic stress disorder, panic disorder, bulimia or anorexia nervosa if previously present, must be in remission for 6 months as defined by DSM-IV-TR criteria, derived from the MINI;
9. Alcohol, medication, or illegal substance dependence within last 12 months;
10. Advanced cardiovascular disease which renders anesthesia and surgery as unsafe as determined by neurosurgeon;
11. Plans to use diathermy;
12. Have any metallic implants in the brain such as aneurysm clips or cochlear implants;
13. Currently participating in another investigational device, drug or surgical trial.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy: Changes in the Hamilton Depression Rating Scale-17 | 3 and 6 months
  evaluate change in HAMD-17 3 months and 6 months after implantation

SECONDARY OUTCOMES:
The incidence of all adverse events | 6 months
  The incidence of all adverse events (i.e. hospitalization due to worsening depression, suicidal ideation, or behavior, medical treatment, and device related events) that occur over study duration.
Showing SCG-DBS significantly increases health related quality of life compared to sham stimulation in patients with TRD | 6 months
  The following health related quality of life measures will be evaluated: Sheehan Disability Scale-Visual Analog Scale (SDS-VAS), Short Form-12 (SF-12), Sexual Functioning questionnaire (SEX FX) and Endicott Work Productivity Scale (EWPS). Each measure will be evaluated at baseline and the after each treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Sidney Kennedy, M.D., Principal Investigator — Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada